CLINICAL TRIAL: NCT00000910
Title: Medical Chart Abstraction of HIV-Infected Pregnant Women and Their Infants Receiving Care or Consultation at Study Sites
Brief Title: A Study to Collect Information About HIV-Positive Pregnant Women and Their Babies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG 367; PACTG 367; 11330 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to collect medical information about HIV-positive pregnant women and their babies who have been (or are being) seen at study sites. This information will be used to help design future research studies for these patients.

The population of HIV-positive pregnant women and their babies who are seen at study sites has not been officially examined. In order to design future studies to research the best care for these patients, this study will examine important characteristics and the general number of women in these trials.

DETAILED DESCRIPTION:
The population served at affiliated ACTG sites has not been officially described. Anecdotal evidence, however, has surfaced regarding the characteristics of HIV-infected pregnant women and the current standard of care during pregnancy. This chart abstraction study is designed to define, more accurately, the pertinent characteristics and general numbers of women in these trials.

In this medical chart abstraction study, pertinent information is collected on all HIV-infected pregnant women and their infants who receive primary or consultative care at PACTG 367 study sites. Part A profiles all HIV-infected women who received care or consultation at study sites and who had a pregnancy outcome between January 1, 1998 through July 1, 1998. [AS PER AMENDMENT 04/12/02: Part A is closed to enrollment.] Part B profiles HIV-infected pregnant women who receive primary or consultative care and a pregnancy outcome following July 1, 1998.

ELIGIBILITY:
Inclusion Criteria

A patient may be eligible for this study if she:

* Is an HIV-positive woman.
* Is receiving care at a study site during the study period or her infant is receiving care at a study site and whose delivery information is available.
* Had a baby on or after January 1, 1998.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Tuomala, Study Chair; Renee Samelson, Study Chair
Locations (2):
- United States (2):
  - Brigham and Women's Hosp., Div. of Infectious Disease, Boston, Massachusetts
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey